CLINICAL TRIAL: NCT06389344
Title: Effect of Esketamine on Conscious State in Patients With Prolonged Disorders of Consciousness#a Prospective, Randomized, Exploratory Study
Brief Title: Effect of Esketamine on Conscious State in Patients With pDoC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lk20240401
Record Dates: First submitted 2024-04-17; First posted 2024-04-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Esketamine; Consciousness Disorders
MeSH Terms: conditions — Consciousness Disorders | interventions — Esketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- esketamine (Experimental): Esketamine ( 50mg, dissolved in 50ml normal saline ) 0.3mg / kg will be infused intravenously at a constant speed within 30 min after tracheal intubation/pneumatectomy fixation.
  Interventions: Drug: Esketamine
- normal saline (Placebo Comparator): Same amount of normal saline will be infused intravenously at a constant speed within 30 min after tracheal intubation/pneumatectomy fixation.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: Esketamine — Esketamine ( 50mg, dissolved in 50ml normal saline ) 0.3mg / kg will be infused intravenously at a constant speed within 30 min after tracheal intubation/pneumatectomy fixation.
  Arms: esketamine
Drug: normal saline — Same amount of normal saline will be infused intravenously at a constant speed within 30 min after tracheal intubation/pneumatectomy fixation.
  Arms: normal saline

SUMMARY:
The goal of this clinical trial is to learn about the effect of intraoperative infusion of subanesthetic dose of esketamine on conscious status in patients with prolonged disorders of consciousness under sevoflurane anesthesia.

Participants will be patients with prolonged disorders of consciousness undergoing surgery with general anesthesia at Beijing Tiantan Hospital. 0.3mg/kg esketamine or saline will be infused will be infused intravenously at a constant speed within 30 min after tracheal intubation/pneumatectomy fixation. Coma recovery scale-revised, Glasgow coma scale, Full Outline of UnResponsiveness scores, SedLine multi-channel electroencephalogram and perioperative adverse events after surgery will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1.16-65 years old 2.Native Chinese language 3.pDoC after acquired brain injury 4.Scheduled to undergo surgery 5.Signed informed consent

Exclusion Criteria:

1. Continuous sedation treatment was carried out within 72 hours before the study
2. Airway stenosis and severe ventilation or ventilation dysfunction caused by various reasons
3. Known or suspected to have serious cardiac, pulmonary and renal dysfunction 1)Severe cardiac dysfunction: a. unstable coronary syndrome b. Congestive heart failure: left ventricular ejection fraction less than 50%, elevated BNP c.Severe arrhythmia d. History of severe valvular disease 2)Severe pulmonary dysfunction: a. history of pulmonary heart disease b. History of chronic obstructive pulmonary disease 3)Severe renal dysfunction: a. Endogenous creatinine clearance (Ccr) less than 30ml/min b. The glomerular filtration rate (GFR) was less than 30ml/min•1.73m2
4. Allergic history of sedative drugs
5. Combined with other mental or nervous system diseases
6. Other reasons are not suitable for this study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Coma recovery scale-revised(CRS-R) | 3±1 day after surgery
  The CRS-R ranges from 0 to 23, with a higher score indicating a better state of consciousness.

SECONDARY OUTCOMES:
Coma recovery scale-revised(CRS-R) | 1,3,6 months after surgery
  The CRS-R ranges from 0 to 23,with a higher score indicating a better state of consciousness.
Full Outline of UnResponsiveness(FOUR) | 3±1 day, 1,3,6 months after surgery
  The FOUR ranges from 0 to 16, with a higher score indicating a better state of consciousness.
Glasgow coma scale(GCS) | 3±1 day, 1,3,6 months after surgery
  The GCS ranges from 3 to 15,with a higher score indicating a better state of consciousness.
Original EEG | during surgery and 3±1 day after surgery
Patient state index(PSI) | during surgery and 3±1 day after surgery
Power spectral density | during surgery and 3±1 day after surgery
Burst-suppression ratio | during surgery and 3±1 day after surgery
Spectral edge frequency | during surgery and 3±1 day after surgery
The incidence of perioperative adverse events | 3±1 day, 1,3,6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China